CLINICAL TRIAL: NCT03351985
Title: the Effect of Quantitative Electroencephalogram (qEEG) in Predictive of Post-operation Delirium and Prognosis of Cardiac Surgery Patients
Brief Title: The Study of Post-operation Delirium and Prognosis of Cardiac Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, professor, Southeast University, China
Other Study IDs: 2017ZDSYLL054-P01
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium Group: The cardiac surgery patients with delirium receive the quantitative electroencephalogram (qEEG) monitoring within 1 hour when they admitted to ICU
  Interventions: Device: quantitative electroencephalogram (qEEG)
- Non-delirium Group: The cardiac surgery patients without delirium receive the quantitative electroencephalogram (qEEG) monitoring within 1 hour when they admitted to ICU
  Interventions: Device: quantitative electroencephalogram (qEEG)

INTERVENTIONS:
Device: quantitative electroencephalogram (qEEG) — the patients receive the quantitative electroencephalogram (qEEG) monitoring within 1 hour when they admitted to ICU

SUMMARY:
Delirium is the most common neurological complication of cardiac surgery patients and associated with poor prognosis. In recent years, the important role of quantitative electroencephalogram (qEEG) in brain function monitoring is becoming increasingly prominent. The purpose of this study is to evaluate the effect of qEEG in predictive of post-operation delirium and prognosis of cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patients of cardiac surgery aged ≥18 years
2. Signed informed consent

Exclusion Criteria:

1. Patients with a history of any neurologic and psychiatric disease
2. Cognitive disorder
3. Stroke history in three years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving cardiac surgery
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
amplitude integrated electroencephalogram (aEEG) | 24 hours
  the electroencephalogram amplitude of cardiac surgery patients assessed by quantitative electroencephalogram when admitted to intensive care unit

SECONDARY OUTCOMES:
alpha frequency band energy | 24 hours
  the percentage of alpha frequency band of cardiac surgery patients assessed by quantitative electroencephalogram when admitted to intensive care unit
beta frequency band energy | 24 hours
  the percentage of beta frequency band of cardiac surgery patients assessed by quantitative electroencephalogram when admitted to intensive care unit
theta frequency band energy | 24 hours
  the percentage of theta frequency band of cardiac surgery patients assessed by quantitative electroencephalogram when admitted to intensive care unit
delta frequency band energy | 24 hours
  the percentage of delta frequency band of cardiac surgery patients assessed by quantitative electroencephalogram when admitted to intensive care unit
alpha variability | 24 hours
  the variability of alpha frequency band of cardiac surgery patients assessed by quantitative electroencephalogram when admitted to intensive care unit
arterial oxygen saturation (SaO2) | 24 hours
  the level of arterial oxygen saturation (SaO2) of cardiac surgery patients when admitted to intensive care unit
central venous oxygen saturation (ScvO2) | 24 hours
  the level of central venous oxygen saturation(ScvO2) of cardiac surgery patients when admitted to intensive care unit
neuron specific enolase (NSE) | 24 hours
  the level of neuron specific enolase (NSE) of cardiac surgery patients when admitted to intensive care unit
interleukin-6 (IL-6) | 24 hours
  the level of interleukin-6 (IL-6) of cardiac surgery patients when admitted to intensive care unit
troponin i (TNI) | 24 hours
  the level of troponin i (TNI) of cardiac surgery patients when admitted to intensive care unit
high-sensitivity C-reactive protein (hs-CRP) | 24 hours
  the level of high-sensitivity C-reactive protein (hs-CRP) of cardiac surgery patients when admitted to intensive care unit
N-terminal pro brain natriuretic peptide (NT-pro-BNP) | 24 hours
  the level of N-terminal pro brain natriuretic peptide (NT-pro-BNP) of cardiac surgery patients when admitted to intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Liu Wenxue, master, Principal Investigator — Southeast University

REFERENCES:
- [Derived] Guo Z, Wan W, Liu W, Liu L, Yang Y, Yang C, Cui X. Quantitative electroencephalography predicts postoperative delirium in adult cardiac surgical patients from a prospective observational study. Sci Rep. 2024 Dec 28;14(1):31101. doi: 10.1038/s41598-024-82422-7. PMID 39730694